CLINICAL TRIAL: NCT01185418
Title: Evaluation of Negative Symptoms and Cognitive Function After Administration of Antipsychotics in Healthy Volunteer: a Double-blind, Randomized Trial of a Single Dose of Placebo, Haloperidol, Amisulpride, Risperidone and Aripiprazole
Brief Title: Evaluation of Negative Symptoms and Cognitive Function After Administration of Antipsychotics in Healthy Volunteer
Status: Completed | Type: Observational
Sponsor: Chonbuk National University Hospital (Other)
Responsible Party: Young Chul Chung/Professor of Psychiatry, Chonbuk National University Hospital, Jeonju, Korea
Other Study IDs: CBIRB0226-22
Record Dates: First submitted 2010-08-18; First posted 2010-08-20 (Estimated); Last update posted 2010-08-20 (Estimated); Status verified 2009-03

CONDITIONS: Normal Volunteers
MeSH Terms: interventions — Risperidone; Aripiprazole; Haloperidol; Amisulpride; Lactose

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- risperidone
  Interventions: Drug: risperidone
- aripiprazole
  Interventions: Drug: aripiprazole
- haloperidol
  Interventions: Drug: haloperidol
- amisulpride
  Interventions: Drug: amisulpride
- lactose
  Interventions: Drug: lactose

INTERVENTIONS:
Drug: risperidone
  Groups: risperidone
Drug: aripiprazole
  Groups: aripiprazole
Drug: haloperidol
  Groups: haloperidol
Drug: amisulpride
  Groups: amisulpride
Drug: lactose
  Groups: lactose

SUMMARY:
The aim of the study is to investigate the negative symptoms and cognitive function after administration of antipsychotics in healthy volunteer.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-38 years and meet no DSM-IV diagnostic criteria as assessed by using the Structured Clinical Interview for DSM-IV, research version.

Exclusion Criteria:

* 1) anyone who participated in other clinical trials within 30 days from the start of this clinical trial or is currently participating in one,
* 2) anyone who has progressive disease or in unstable medical condition unfit for the trial,
* 3) anyone who has been diagnosed in psychiatric terms in the past, depends on psychotropic substance, or has overdosed or depended on the substance or alcohol (except for coffee or tobacco) within 1 month from the trial start,
* 4) anyone who is suicidal or highly probable of suicides, or
* 5) anyone who has test results considered clinically meaningful

Ages: 18 Years to 38 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Recruited volunteers among normal adults aged from 18 to 38 who responded advertisements for research subjects. Then selected subjects from the applicants using various screening tests - physical and neurological examination including confirming vital signs after examining physical health and sleep habits of volunteers
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2009-03; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Symptoms assessment by objective and subjective rating scale | 2 hour
  VAS - mental sedation (alert-drowsy, muzzy-clear headed, mentally slow-quick witted, attentive-dreamy), physical sedation (strong-feeble, well coordinated-clumsy, lethargic-energetic, incompetent-proficient), tranquilization (calm-excited, contented-discontented, troubled-tranquil, tense-relaxed)
Symptoms assessment by objective and subjective rating scales & CNT | 4hour
  SANS-alogia and blunted affect, SDSS-Subjective Deficit Syndrome Scale ,self-report questionnaire to measure lack of energy, blunted affect, and difficulty in or altered thinking, consisting of 19 questions, with the scales from 0 to 4 NIDSS-consists of 20 items with a five-point Likert scale (from 0, none to 4, severe) and has three subscales: avolition (five items), blunted affect (five items), and cognition (ten items), CNT-computerized neuropsychological test, VAS
Symptoms assessment by objective and subjective rating scales | 24hour
  SANS, SDSS, NIDSS, VAS SANS-alogia and blunted affect, SDSS-Subjective Deficit Syndrome Scale ,self-report questionnaire to measure lack of energy, blunted affect, and difficulty in or altered thinking, consisting of 19 questions, with the scales from 0 to 4 NIDSS-consists of 20 items with a five-point Likert scale (from 0, none to 4, severe) and has three subscales: avolition (five items), blunted affect (five items), and cognition (ten items), VAS

SECONDARY OUTCOMES:
Symptoms assessment by objective rating scale | 4hour
  BARS-Barnes akathisia rating scale (BAS), consisting of 4 items, identifies drug-induced akathisia and measures severity, SAS-Simpson-angus scale (SAS), consisting of 10 items, measures neuroleptic induced parkinsonism
Symptoms assessment by objective rating scale | 24hour
  BARS, SAS

CONTACTS AND LOCATIONS:
Locations (1):
- Chonbuk national university hospital, Jeonju, South Korea